CLINICAL TRIAL: NCT07222501
Title: Comprehensive Self-Management Support for WTC Responders With Asthma
Brief Title: NIOSH R21 WTC Asthma
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Juan Wisnivesky, Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 23-2262
Record Dates: First submitted 2025-10-27; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Asthma Education - WTC Related: 1-3 visits with an asthma educator to receive basic asthma education. The number and times of the meetings will be determined by the participant.
  Interventions: Behavioral: Asthma Education - WTC Related
- Self Management Support with Lay Health Coaches: Supporting Self-Management Behaviors for Adults (SaMBA) program. The SaMBA model of SMS is an evidence-based approach grounded in a theory of health behavior, the Self-regulation Model (SRM), and a conceptual model of health care use, the Aday-Anderson model. SaMBA is unique among chronic illness SMS programs because its strategy involves comprehensively screening for barriers to effective self-management and disease control and couples it with tailored, theory-based, barrier specific interventions.
  Interventions: Behavioral: SaMBA

INTERVENTIONS:
Behavioral: SaMBA — The health coach will ask many questions to determine how best to help asthma management and to improve asthma control. The intervention lasts 3 months. During those 3 months, the health coach will speak with participant by phone or video chat several times. Meetings will occur once a week for the first 2-3 weeks, then every 2-4 weeks until the intervention ends. The days and times of the meetings will be up to the participant.
  Other Names: Supporting Self-Management Behaviors for Adults
  Groups: Self Management Support with Lay Health Coaches
Behavioral: Asthma Education - WTC Related — 1-3 visits with an asthma educator to receive basic asthma education
  Groups: Asthma Education - WTC Related

SUMMARY:
Aim 2: Conduct a pilot RCT of SaMBA-WTC to determine feasibility and preliminary impact in preparation for a fully powered trial. (7M-24M) The investigators will conduct a pilot RCT (n=58) of the SaMBA-WTC model vs. an attention control. Data will be collected on the primary outcomes (asthma control [asthma control test, ACT], medication use, inhaler technique) as well as on other secondary outcomes including measures of physical function, self-management behaviors, feasibility and fidelity at baseline, at intervention completion at 3 months, and for sustainability at 6 months. This project will prepare the team for all aspects of a subsequent larger efficacy trial of SaMBA-WTC.

ELIGIBILITY:
Inclusion Criteria:

* Age >=21 years;
* English or Spanish speaking;
* World Trade Center-certified asthma;
* on asthma controller medications (as needed or standing);
* uncontrolled asthma.

Exclusion Criteria:

* Physician's diagnosis of dementia,
* COPD or other chronic pulmonary disease,
* >15 pack-years history of smoking to avoid enrolling WTC responders with undiagnosed COPD.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: World Trade Center Responders from the World Trade Center Health Program at Mount Sinai
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) | 12 months and 3 months post intervention
  Asthma control test assesses how well asthma is controlled over the past four weeks. Total score range from 5-25, with higher score indicating better health outcomes.
Number of times controller inhaler used | 12 months and 3 months post intervention
  Medication use will be measured with electronic monitors attached to the participant's control inhaler. Adherence will be measured by use of the electronic monitors that will capture how often the participant uses their controller inhaler.

SECONDARY OUTCOMES:
Mini Asthma Quality of Life Questionnaire (AQLQ) | 12 months and 3 months post intervention
  The validated Mini Asthma Quality of Life Questionnaire (AQLQ) is available in English and Spanish. The 15-item questionnaire measures quality of life in the domains of symptoms, activity limitation, emotional function, and environmental stimuli. Items are scored on a 7-point scale from severely impaired to not impaired at all. Each domain scores and full scores range 1-7, with higher scores indicating better quality of life.
Number of Hospital visits | 12 months and 3 months post intervention
  Any hospital visits at every research visit will be track by use of survey in REDCap.
Number of Emergency Department visits | 12 months and 3 months post intervention
  Any emergency visits at every research visit will be track by use of survey in REDCap.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Wisnivesky, MD, DrPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Proposals should be directed to juan.wisnivesky@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link tbd).